CLINICAL TRIAL: NCT00617019
Title: A Cross-sectional, Retrospective Screening and Case-control Study Examining the Frequency of, and Risk Factors Associated With, Impulse Control Disorders in Parkinson's Disease Patients Treated With MIRAPEX® (Pramipexole) and Other Anti-parkinson Agents (DOMINION Study)
Brief Title: Impulse Control Disorders in Parkinson's Patients Treated With Pramipexole and Other Agents (DOMINION Study)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 248.619; DOMINION
Record Dates: First submitted 2008-02-05; First posted 2008-02-15 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Parkinson's patients: Observational study to compare rates of impulse control disorders in patients taking different medications for Parkinson's Disease

SUMMARY:
The purpose is to explore the frequency of impulse control disorders in Parkinson's patients treated with different Parkinson's medications.

ELIGIBILITY:
Inclusion Criteria:

Observation Criteria:

Male or female outpatients, aged 30 to 75 years of age, with idiopathic PD. Patients must be selected on the basis of a prospective recruitment plan documented at the site, with the objective of obtaining an unbiased representative sample.

Patients must have been treated with anti-parkinson medication for a period of one year or greater and demonstrated a treatment response, in the opinion of the Investigator.

Patients must be willing and able to comply with study procedures. Patients must be willing and able to give meaningful, written informed consent. This must be completed prior to beginning any study procedures, in accordance with GCP and local legislation.

Exclusion Criteria:

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson's patients treated with various medications
Sampling Method: Non-Probability Sample
Enrollment: 3234 (Actual)
Dates: Start 2006-09; Primary Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of current ImpulseControl Disorder(ICD) assessed via + res. of Modif.Massachusetts Gambling Screen,Modif.Minnesota Impulsive Disorder Interview for Sexuality,Modif.MIDI for Compulsive Buying,DSM-IV binge-eating research criteria questionnaire | 6 months

SECONDARY OUTCOMES:
The occurrence of a past (since onset of PD) ICD | 6 months
Demographic and medical history measures | up to 14 days after Visit 1
Scores on psychiatric/neuropsychological instruments/tests | up to 14 days after Visit 1

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (49):
- United States (36):
  - 248.619.01034 Neurological Physicians of Arizona, Gilbert, Arizona
  - 248.619.01007 Mayo Clinic - Scottsdale, Scottsdale, Arizona
  - 248.619.01025 Sun Health Research Institute, Sun City, Arizona
  - 248.619.01018 Margolin Brain Institute, Fresno, California
  - 248.619.01031 Pacific Neuroscience Medical Group, Inc., Oxnard, California
  - 248.619.01016 San Francisco VA PD Research, Education, & Clinical Center, San Francisco, California
  - 248.619.01023 The Parkinson's Institute, Sunnyvale, California
  - 248.619.01021 Boehringer Ingelheim Investigational Site, Englewood, Colorado
  - 248.619.01027 Associated Neurologists, P.C., Danbury, Connecticut
  - 248.619.01013 Molecular NeuroImaging, New Haven, Connecticut
  - 248.619.01020 Parkinson's Disease and Movement Disorders of Boca Raton, Boca Raton, Florida
  - 248.619.01009 University of Florida, Gainesville, Florida
  - 248.619.01035 Emory University, Atlanta, Georgia
  - 248.619.01006 Medical College of Georgia, Augusta, Georgia
  - 248.619.01014 Northwestern University, Chicago, Illinois
  - 248.619.01001 The University of Kansas Medical Center, Kansas City, Kansas
  - 248.619.01015 John Hopkins Hospital, Baltimore, Maryland
  - 248.619.01029 Clinical Neuroscience Center, Southfield, Michigan
  - 248.619.01022 University of Minnesota, Minneapolis, Minnesota
  - 248.619.01008 Robert Wood Johnson Medical School, Piscataway, New Jersey
  - 248.619.01030 Parkinson's Disease and Movement Disorders Center, Albany, New York
  - 248.619.01036 Parkinson's Disease and Mov. Disorders Center of Long Island, Commack, New York
  - 248.619.01017 Weill Cornell medical College, New York, New York
  - 248.619.01003 Duke University Medical Center, Durham, North Carolina
  - 248.619.01028 The Cleveland Clinic Foundation, Cleveland, Ohio
  - 248.619.01004 Lehigh Valley Hospital, Allentown, Pennsylvania
  - 248.619.01010 Parkinson's Disease research, Education and Clinical Center, Philadelphia, Pennsylvania
  - 248.619.01011 University of Pennsylvania, Philadelphia, Pennsylvania
  - 248.619.01024 Thomas Jefferson Hospital, Philadelphia, Pennsylvania
  - 248.619.01019 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 248.619.01012 Parkinson's Disease and Movement Disorders Center, Upland, Pennsylvania
  - 248.619.01005 NeuroHealth, Warwick, Rhode Island
  - 248.619.01033 Vanderbilt University Medical Center, Nashville, Tennessee
  - 248.619.01032 Neurology Spclst of Dallas, PA, Dallas, Texas
  - 248.619.01002 Baylor College of Medicine, Houston, Texas
  - 248.619.01026 Neurology/Southeast Parkinson's Disease, Richmond, Virginia
- Canada (13):
  - 248.619.02011 University of Calgary, Calgary, Alberta
  - 248.619.02010 The Glenrose Rehab. Hospital, Edmonton, Alberta
  - 248.619.02009 Movement Disorder Clinic, Winnipeg, Manitoba
  - 248.619.02005 Health Sciences Centre, St. John's, Newfoundland and Labrador
  - 248.619.02019 Dr. David King, Halifax, Nova Scotia
  - 248.619.02013, Kitchener, Ontario
  - 248.619.02018 London HSC - University Hospital, London, Ontario
  - 248.619.02001 Centre for Movement Discorder, Markham, Ontario
  - 248.619.02008 Ottawa Civic Hospital, Ottawa, Ontario
  - 248.619.02016 The Toronto Western Hospital, Toronto, Ontario
  - 248.619.02003 Unite des Troubles du Mouvement, Montreal, Quebec
  - 248.619.02002 Memory and Motor Skills Disorders Clinic, Québec, Quebec
  - 248.619.02017 Royal University Hospital, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Weintraub D, Koester J, Potenza MN, Siderowf AD, Stacy M, Voon V, Whetteckey J, Wunderlich GR, Lang AE. Impulse control disorders in Parkinson disease: a cross-sectional study of 3090 patients. Arch Neurol. 2010 May;67(5):589-95. doi: 10.1001/archneurol.2010.65. PMID 20457959